CLINICAL TRIAL: NCT00584194
Title: Parts A&B: Evaluation of the Safety and Immunogenicity of Rift Valley Fever Vaccine, Inactivated, Dried (TSI-GSD 200), A Phase 2 Study
Brief Title: Safety and Immunogenicity Study of Rift Valley Fever Vaccine
Acronym: RVF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A-12592; FY03-05 (Other: SIP)
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Rift Valley Fever
Keywords: Hemorrhagic Fever, Viral Infections, Neurologic diseases, Arbovirus Infections, RVF
MeSH Terms: conditions — Rift Valley Fever; Hemorrhagic Fevers, Viral; Virus Diseases; Nervous System Diseases; Arbovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TSI-GSD 200 RVF Vaccine (Experimental): Part A: Inactivated, Dried (TSI-GSD 200) RVF vaccine, will be given as three 1.0-ml subcutaneous primary series injections, with doses on day 0, once on days 7-14, once on days 28-42 (the third dose will be given at least 21 days after the second dose).Part B: Subcutaneous 1.0-ml booster doses (maximum of four boosters over 12 months) will be given if the volunteer fails to respond to the primary series with a PRNT80 ≥ 1:40 or annually if titer wanes to < 1:40.
  Interventions: Biological: TSI-GSD 200 RVF Vaccine

INTERVENTIONS:
Biological: TSI-GSD 200 RVF Vaccine — Part A: Inactivated, Dried (TSI-GSD 200) RVF vaccine will be given as three 1.0-ml subcutaneous primary series injections, with doses on day 0, once on days 7-14, once on days 28-42 (the third dose will be given at least 21 days after the second dose).Part B: Subcutaneous 1.0-ml booster doses (maximum of four boosters over 12 months) will be given if the volunteer fails to respond to the primary series with a PRNT80 ≥ 1:40 or annually if titer wanes to < 1:40.

SUMMARY:
This study is designed to determine the safety and immunogenicity of a Rift Valley Fever (RVF) Vaccine

DETAILED DESCRIPTION:
Study Objectives:

The objectives of this two-part, primary immunization and booster dose, study are to continue to collect safety data on Rift Valley Fever (RVF) Vaccine, Inactivated (TSI-GSD 200); and, to continue to collect immunogenicity data on Rift Valley Fever (RVF) Vaccine, Inactivated (TSI-GSD 200) and analyze interim data to determine whether a 6-month dose is indicated; and, to provide potential protection for personnel at risk for occupational exposure to the RVF virus and collect data on incidence of occupational RVF infection (subclinical and clinical) in immunized personnel.

ELIGIBILITY:
Inclusion Criteria:

Parts A & B:

* At least 18 years old, or if active military duty, 17 years old,
* Females of childbearing potential must agree to have a urine pregnancy test within 48 hours before receipt of each dose of vaccine. The test results must be negative. Females will be advised not to become pregnant for 3 months after the primary series and each booster dose, and must not be breast-feeding,
* Subject must be actively enrolled in the SIP to be vaccinated at USAMRIID or be otherwise authorized (with documentation) by the DOD
* Subjects must be at risk for exposure to RVF virus,
* Subjects must have an up-to-date (within 1 year) medical history, physical examination, and laboratory tests in their charts and be medically cleared for participation by an investigator. Examinations or tests may be repeated within 1 year at the discretion of the enrolling physician.
* Volunteer must have signed and dated the approved informed consent (Volunteer Agreement Explanation and Affidavit).

Additional Inclusion Criteria for Part B:

• Completion of primary series and any follow-up titer (PRNT80) < 1:40 from the current or a previous RVF IND 365 protocol.

Exclusion Criteria

Parts A & B:

* Clinically significant abnormal lab results including evidence of Hepatitis C, Hepatitis B or carrier state, or elevated liver function tests.
* Personal history of immunodeficiency or current treatment with immunosuppressive medication, at the discretion of the physician.
* Confirmed HIV infection.
* Any medical condition that, at the discretion of the physician, may jeopardize the safety of the volunteer.
* Any serious or life-threatening allergies to any component of the vaccine: formalin, human serum albumin, neomycin, streptomycin
* Administration of any other vaccine within 28 days of any dose of RVF vaccine.
* Any unresolved adverse event resulting from a previous immunization.

Additional Exclusion Criteria for Part B:

• An adequate PRNT80 (≥ 1:40) after completion of primary series.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2004-06 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Rusnak, MD, Principal Investigator — USAMRIID Medical Division
Locations (1):
- U.S. Army Medical Research Institute of Infectious Diseases, Fort Deterick, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 278 subjects were enrolled at USAMRIID to participate
Period: Overall Study
Arm/Group | TSI-GSD 200 RVF Vaccine
Started | 278
Completed | 143
Not Completed | 135
Not completed — Other | 135

BASELINE CHARACTERISTICS:
Population: Baseline includes all subjects vaccinated and doesn't account for drop outs, deviations, and withdraws. Demographics weren't given in Final Clinical Study Report. Numbers are reliant on numbers of females and males receiving vaccination.
Arm/Group | TSI-GSD 200 RVF Vaccine
Number analyzed (Participants) | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 153
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 103
Region of Enrollment [Number; unit: participants]
  United States | 153

OUTCOME MEASURES:

1. Primary Outcome: Safety: All Incidences of Erythema
Description: Collect data on the occurrence of AEs and SAEs in reference to Erythema (most frequently reported AE) in parts A and B of the study
Time Frame: 12 months
Measure: Number; unit: number of events
Arm/Group | TSI-GSD 200 RVF Vaccine
Number analyzed (Participants) | 278
number of events
  Mild | 15
  Moderate | 10
  Severe | 0

2. Secondary Outcome: Immunogenicity: Geometric Mean Titers After 3rd Vaccination
Description: Measurement is the 80% plaque-reduction neutralization titer (PRNT80) antibodies to RVF virus following 3rd vaccination (Parts A and B of study)
Time Frame: 28 days after dose 3
Population: Population is based on responders (defined as a subject achieving a PRNT80 >1:40)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TSI-GSD 200 RVF Vaccine
Number analyzed (Participants) | 102
Titers
  Male: GMT | 47.3 [29.6 to 75.4]
  Female: GMT | 74.9 [43.6 to 128.6]

3. Secondary Outcome: Immunogenicity: Geometric Mean Titers Before 6-month Booster
Description: Measurement is the 80% plaque-reduction neutralization titer (PRNT80) for study Parts A and B
Time Frame: Before 6-month booster
Population: Population is based on responders (defined as a subject achieving a PRNT80 >1:40)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TSI-GSD 200 RVF Vaccine
Number analyzed (Participants) | 39
Titers
  Male: GMT | 8.5 [4.7 to 15.3]
  Female: GMT | 23.9 [8.2 to 68.9]

4. Secondary Outcome: Immunogenicity: Geometric Mean Titers at 12 Months
Description: Measurement is the 80% plaque-reduction neutralization titer (PRNT80) for study Parts A and B.
Time Frame: at 12 months
Population: Population is based on responders (defined as a subject achieving a PRNT80 >1:40)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TSI-GSD 200 RVF Vaccine
Number analyzed (Participants) | 24
Titers
  Male: GMT | 48.8 [20.1 to 118.1]
  Female: GMT | 48.4 [23.1 to 101.5]

5. Secondary Outcome: Immunogenicity: Geometric Mean Titers After 6-month Booster
Description: Measurement is the 80% plaque-reduction neutralization titer (PRNT80) for study Parts A and B.
Time Frame: month 6 after dose 4
Population: Population is based on responders (defined as a subject achieving a PRNT80 >1:40)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TSI-GSD 200 RVF Vaccine
Number analyzed (Participants) | 67
Titers
  Male: GMT | 211.8 [140.5 to 319.3]
  Female: GMT | 189.0 [128.0 to 279.0]

ADVERSE EVENTS:
Time Frame: Annuals done for 5 years
Description: Of the 278 subjects enrolled, 153 subjects received at least 1 vaccination of Rift Valley Fever Vaccine, Inactivated, Dried (TSI-GSD 200) and 125 subjects were enrolled in the study but did not receive RVF vaccine. Each dose (primary, booster, or supplemental) consisted of 1.0 mL of vaccine delivered subcutaneously in the upper outer aspect of the arm (triceps area).
Arm/Group | TSI-GSD 200 RVF Vaccine
All-Cause Mortality (participants affected / at risk) | 0/153
Serious Adverse Events (participants affected / at risk) | 11/153
Other Adverse Events (participants affected / at risk) | 75/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TSI-GSD 200 RVF Vaccine (N=153)
Rotator cuff surgery (Surgical and medical procedures) | 1 (1)
Cyst exicision (Skin and subcutaneous tissue disorders) | 1 (1)
Loss of consciousness during physcial assault (Injury, poisoning and procedural complications) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 1 (1)
Obstructive sleep apnea surgery (Surgical and medical procedures) | 1 (1)
Back surgery (Surgical and medical procedures) | 1 (1)
Meniscus repair surgery (Surgical and medical procedures) | 1 (1)
Partial sigmoidectomy (Surgical and medical procedures) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Laproscopic surgery for RLQ pain (Surgical and medical procedures) | 1 (1)
Left nephrectomy (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TSI-GSD 200 RVF Vaccine (N=153)
Headache (Nervous system disorders) | 1 (1) — Unrelated
Headache (Nervous system disorders) | 13 (13) — Possibly related
Headache (Nervous system disorders) | 1 (1) — Unlikely related
Headache (Nervous system disorders) | 2 (2) — Probably related
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) — Definitely related
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) — Unrelated
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) — Unlikely related
Fatigue (General disorders) | 2 (2) — Unrelated
Fatigue (General disorders) | 8 (8) — Possibly related
Fatigue (General disorders) | 1 (1) — Unlikely related
Sore throat (Gastrointestinal disorders) | 3 (3) — Unrelated
Sore throat (Gastrointestinal disorders) | 2 (2) — Possibly related
Sore throat (Gastrointestinal disorders) | 4 (4) — Unlikely related
Malaise (General disorders) | 2 (2) — Unrelated
Malaise (General disorders) | 6 (6) — Possibly related
Malaise (General disorders) | 1 (1) — Unlikely related
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) — Possibly related
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Unlikely related
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) — Unrelated
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Possibly related
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unlikely related
Bruising (Injury, poisoning and procedural complications) | 1 (1) — Unrelated
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) — Possibly related
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unlikely related
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Unrelated
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Possibly related
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unlikely related
Nausea (Gastrointestinal disorders) | 1 (1) — Unrelated
Nausea (Gastrointestinal disorders) | 2 (2) — Possibly related
Nausea (Gastrointestinal disorders) | 2 (2) — Unlikely related
Chills (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Chills (Musculoskeletal and connective tissue disorders) | 2 (2) — Possibly related
Chills (Musculoskeletal and connective tissue disorders) | 1 (1) — Unlikely related
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Unrelated
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Possibly related
Fever (General disorders) | 1 (1) — Unrelated
Fever (General disorders) | 2 (2) — Possibly related
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Possibly related
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unlikely related
Diarrhea (Gastrointestinal disorders) | 2 (2) — Unlikely related
Stuffy nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Stuffy nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unlikely related
warm (General disorders) | 1 (1) — Unlikely related
Fracture (Injury, poisoning and procedural complications) | 2 (2) — Unrelated
Lacerations (Injury, poisoning and procedural complications) | 2 (2) — Unrelated
Pain (General disorders) | 2 (2) — Unrelated
Axillary tenderness (General disorders) | 1 (1) — Definitely related
Swelling (General disorders) | 1 (1) — Unlikely related
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related
Chest pain (Cardiac disorders) | 1 (1) — Unrelated
Chest pain (Cardiac disorders) | 1 (1) — Unlikely related
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unlikely related
Light headedness (Nervous system disorders) | 1 (1) — Unrelated
Light headedness (Nervous system disorders) | 1 (1) — Possibly related
Rash (Skin and subcutaneous tissue disorders) | 2 (2) — Unrelated
Low back pain (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Possibly related
Scratchy throat (Gastrointestinal disorders) | 2 (2) — Possibly related
Abdominal cramping (Gastrointestinal disorders) | 1 (1) — Unlikely related
Head cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unlikely related
Swollen neck glands (Blood and lymphatic system disorders) | 1 (1) — Unrelated
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unlikely related
Admittance (Injury, poisoning and procedural complications) | 1 (1) — Unrelated
Blurred vision (Nervous system disorders) | 1 (1) — Unrelated
Concussion (Injury, poisoning and procedural complications) | 1 (1) — Unrelated
Hives (Immune system disorders) | 1 (1) — Unlikely related
Stomach ache (Gastrointestinal disorders) | 1 (1) — Unlikely related
Foggy head (Nervous system disorders) | 1 (1) — Unrelated
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related
Neck swollen (General disorders) | 1 (1) — Unrelated
Bump on right arm (Injury, poisoning and procedural complications) | 1 (1) — Unrelated
Chest congestion (Infections and infestations) | 1 (1) — Unrelated
Feeling faint (Nervous system disorders) | 1 (1) — Definitely related
Stiff neck (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related
Hoarseness (Psychiatric disorders) | 1 (1) — Unlikely related
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) — Unlikely related
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) — Unlikely related
Tender lymph nodes (Blood and lymphatic system disorders) | 1 (1) — Unlikely related
Tight chest (Cardiac disorders) | 1 (1) — Unlikely related
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unlikely related
Flashes of light (Nervous system disorders) | 1 (1) — Unlikely related
GI problems (Gastrointestinal disorders) | 1 (1) — Unlikely related
Knee injury (Injury, poisoning and procedural complications) | 1 (1) — Unrelated
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Absence from work (General disorders) | 1 (1) — No data
Pressure (General disorders) | 1 (1) — Possibly related
Sinus headache (Nervous system disorders) | 1 (1) — Possibly related
Stomach virus (Gastrointestinal disorders) | 1 (1) — Unrelated
Urination discomfort (Renal and urinary disorders) | 1 (1) — Unrelated
Ear pressure (Ear and labyrinth disorders) | 1 (1) — Unrelated
Bronchitis (Infections and infestations) | 1 (1) — Unrelated
Nail fungus (Infections and infestations) | 1 (1) — Unrelated
Upper eyelid pain to touch (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Upper eyelid itchy (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Upper eyelid swollen (Immune system disorders) | 1 (1) — Unrelated
Muscle strain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Rotator cuff screw removal (Surgical and medical procedures) | 1 (1) — Unrelated
Sweating (General disorders) | 1 (1) — Possibly related
Bradycardia (Cardiac disorders) | 1 (1) — Unrelated
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related
Pinkeye (Infections and infestations) | 1 (1) — Unrelated
Migraine (Nervous system disorders) | 1 (1) — Possibly related
Itchy bumps on arms (Injury, poisoning and procedural complications) | 1 (1) — Probably related
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related
Eye trauma (Injury, poisoning and procedural complications) | 1 (1) — Unrelated
Abcess (Infections and infestations) | 1 (1) — Unrelated
Abdomen pain (Gastrointestinal disorders) | 1 (1) — Unrelated
Bil umbilial hernias (Gastrointestinal disorders) | 1 (1) — Unrelated
Inguinal hernia (Gastrointestinal disorders) | 1 (1) — Unrelated
Face swelling (Immune system disorders) | 1 (1) — Unlikely related
Elevated B/P (Investigations) | 1 (1) — Definitely related
URI (Investigations) | 1 (1) — Possibly related
Pruritus (Skin and subcutaneous tissue disorders) | 11 (11) — Definitely related
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Erythema (Skin and subcutaneous tissue disorders) | 14 (14) — Definitely related
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) — Unrelated
Induration (General disorders) | 10 (10) — Definitely related
Induration (General disorders) | 1 (1) — Unrelated
Tender at site (Injury, poisoning and procedural complications) | 8 (8) — Definitely related
Bruising (Injury, poisoning and procedural complications) | 6 (6) — Definitely related
Warmth at site (Injury, poisoning and procedural complications) | 4 (4) — Definitely related
Tenderness (Injury, poisoning and procedural complications) | 3 (3) — Definitely related
Soreness (Injury, poisoning and procedural complications) | 2 (2) — Definitely related
Warm (General disorders) | 1 (1) — Definitely related
Axillary pain (General disorders) | 1 (1) — Probably related
Swelling (General disorders) | 1 (1) — Definitely related
Edema (Metabolism and nutrition disorders) | 2 (2) — Definitely related
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) — Definitely related
Hot at site (Injury, poisoning and procedural complications) | 1 (1) — Definitely related
Redness (Skin and subcutaneous tissue disorders) | 1 (1) — Definitely related
Burning and pinching (General disorders) | 1 (1) — Unrelated
Tender to touch (Injury, poisoning and procedural complications) | 1 (1) — Definitely related
Burning sensation (Nervous system disorders) | 1 (1) — Definitely related
Pain at site (Injury, poisoning and procedural complications) | 1 (1) — Definitely related
Tingling (Nervous system disorders) | 1 (1) — Definitely related
Swelling at site (Injury, poisoning and procedural complications) | 1 (1) — Definitely related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No